CLINICAL TRIAL: NCT04951440
Title: Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Trial to Evaluate the Effectiveness and Safety of Nitrone for Injection in Patients With Acute Ischemic Stroke
Brief Title: Study on the Effectiveness and Safety of Nitrone for Injection in Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2019009
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Nitroxazine
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: 30min intravenous point. Infusion of 1400 mg of tetranitrone was given to bed I with a dose of 100ml, twice a day, with an interval of 12 hours, and continued administration for 7 days, that is, a total of about 14 times.
  version
  Interventions: Drug: Nitrate ketone oxazine
- Placebo group (Placebo Comparator): Placebo group: 30 minutes to earn pulse, I, 1, and dripping Yunmi gave 100mL placebo (sodium chloride injection). It is administered twice a day for 1 to 2 hours, and the pattern is transferred to about 7 people, that is, about 14 times in total.
  Interventions: Drug: Nitrate ketone oxazine

INTERVENTIONS:
Drug: Nitrate ketone oxazine — Intervention group: 30min intravenous point. Drop qiu was given 1400 mg of injected sichuan nitrone I bed, and the drug was given 100 mL at day F Set 12 h, and at odds with another 7 days, that is, about 14 times in total.

SUMMARY:
The main purpose of the study: To evaluate the effect of nitrosone 1 special for patients with acute ischemic cerebral stroke. The secondary purpose of the study: To evaluate the effectiveness of the injection of nitrosone I. T for loyal patients with acute ischemic stroke All women think.

DETAILED DESCRIPTION:
The main purpose of the study: To evaluate the effect of nitrosone 1 special for patients with acute ischemic cerebral stroke. The secondary purpose of the study: To evaluate the effectiveness of the injection of nitrosone I. T for loyal patients with acute ischemic stroke All women think.

This experiment adopts randomized, double-blind, placebo-controlled parallel design. In patients with acute, ischemic cerebral rate as the research object, after selected exclusion standard screening, if doesn't fit or don't agree with thrombolysis subjects, giving from connect to test a drug or a placebo treatment, if appropriate and agreed to thrombolysis of the subjects with an experimental drug or placebo after thrombolysis treatment.Intervention group: 30) min uniform given 1400 mg intravenous drip injection with ketone wordy, nitrate dosing volume 100 ml. Day delivery, two intervals of 12 h, for seven days in a row, namely to 14 times in total.The placebo group: 30 min to 100 ml placebo at a constant speed intravenous drip (sodium chloride injection), dosing W times a day, 12 h, for seven days in a row, namely to 14 times in total.During treatment, participants in the group after injection with nitrate ketone oxazine (giving injections with nitrate ketone oxazine time window < 6 h, that is, from "the last look normal time" to start infusion nitrate obviously time) or placebo and other foundation treatment. Record for the first time to give the time of nitrate ketone oxazine or placebo for injection, lie between 8 and 12 h 2 times to medicine."After 12 h dosing interval, until finish to 14 times (for convenient subjects out of the hospital and acceptable to 13).Allow this study drug and placebo and thrombolysis drug dosing dual channel at the same timeStop to test drug or placebo, in the group of 8 days, 14 days, 30 days, the 90th day to evaluate curative effect, respectively.In the I the ili is not ah into subgroups according to try tii statistical treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) the age 18 to 65 years of age, gender not limited (including 18 and 65 years old) :(2) according to the Chinese guide of diagnosis and treatment of acute ischemic stroke (2018) with a diagnosis of acute ischemic strokeThe lender;(3) from the "look" normal time to start infusion for lamictal nitrate or placebo < 6 hours, to wake up or stroke due to accurately obtain aphasia, disturbance of consciousness and other symptom onset time, shall be made in patients with the last performance of normal time I;(4) after the first or the last disease incidence after the more good (mkS score 0-1) disease patients again;(5) at the four points < NIHISS score < 24 points;(6) from beginning to the last delivery signed informed consent is willing to take effective contraceptive measures within 6 months after:Understand and abide by the research process and voluntary participation, and sign the informed consent form (informed consent signed by the person or legal representative voluntary).

Exclusion Criteria:

* (1) the patients with recurrent cerebral infarction incidence before mRS score > 1;(2) unconsciousness (NIHSS score la 22 points);(3) neural imaging examination (CT/MRI) suggests intracerebral hemorrhagic disease (such as: hemorrhagic cerebral apoplexy, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.)(4) imaging examination showed middle cerebral artery infarction area > one-third, or ASPECT score < 7 points:(5) transient ischemic attack (TIA) :(6) to prepare or have lines endovascular treatment of patients;(7), severe renal insufficiency: creatinine clearance < 30 mL/min (Cockcroft - Gault formula), blood urea nitrogen and/or muscle > 1.5 times the upper limit of normal value, or other serious kidney function is not complete disease known;Severe liver function damage (8) : ALT, AST > 1.5 times the upper limit of normal value, or other known liver diseases such as acute or chronic hepatitis, liver cirrhosis, etc;(9) hospital routine blood tip: white blood cells < normal lower limit; Hemoglobin < normal lower limit; Hospital to check blood sugar < 2.8 tendency for L, or > 16.8 mmo / /; Temperature > 38 c; Other laboratory examination with clinical significance is unusual, and the researchers of decision should not be set;(10) are poorly controlled hypertension, systolic blood pressure > 220 MMHG 2 120 MMHG and/or diastolic blood pressure:(11) heart rate < 40 times/min and/or heart rate > 120 times/min: nearly six months or line of interventional therapy of acute myocardial infarction (ami), patients with heart failure (in the patients with NYHA class for 111-1 v);(12) in patients with epilepsy: merging other patients with mental illness to cooperation or unwilling to cooperation; Patients with dementia.(13) of malignant tumor, blood, digestive serious illness, or other system.(14) on experimental drug or similar components or materials used for imaging examination allergies;(15) blood positie pregnancy, pregnancy and lactation women:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with NIHSS ≤1 or a reduction of 4 or more points from baseline | On the 14th day of treatment
  Percentage of patients with NIHSS ≤1 or a reduction of 4 or more points from baseline at day 14 of treatment

SECONDARY OUTCOMES:
The change of MRS score | 30th day and the 90th day of treatment
  The change of MRS score (change detection and rate of change) at the 30th day and the 90th day of treatment compared with the plexus line.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Study Chair — Tiantan Hospital, Capital Medical University
Locations (2):
- China (2):
  - : Beijing Dan's self technology co., LTD., Beijing
  - Tiantan Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No